CLINICAL TRIAL: NCT05674864
Title: Effect of Probiotics on Eradication Rate in Patient With Persistent Helicobacter Pylori Infection
Brief Title: Effect of Probiotics on Eradication of Persistent H.Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Noura Elsayed Ahmed Elsaka, Principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Probiotics effect on H.Pylori
Record Dates: First submitted 2022-11-22; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Persistent Helicobacter Pylori Infection
Keywords: probiotics; Persistent Helicobacter Pylori Infection
MeSH Terms: interventions — Lacteol

STUDY DESIGN:
Intervention Model Description: 92 patients with persistent H. pylori infection will be recruited randomly to one of the following groups:
  * Group 1 (Control Group): consists of 46 patients who will receive Amoxicillin 1 gm T.I.D + Lansoprazole 30 mg T.I.D. + Placebo 1 capsule T.I.D for 14 days.
  * Group 2 (Linex ® group): consists of 46 patients who will receive Amoxicillin 1 gm T.I.D + Lansoprazole 30 mg T.I.D + Linex ® capsule (which contains Bifidobacterium Infants, Enterococcus Feacium and Lactobacillus Acidophilus) 1 capsule T.I.D for 14 days.
Who Masked: Participant, Investigator
Masking Description: Blindness will be maintained by the similarity in shape and the appearance of both the Linex ® capsule and placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Control Group) (Placebo Comparator): consists of 46 patients who will receive Amoxicillin 1 gm three times daily plus Lansoprazole 30 mg three times daily plus Placebo 1 capsule three times daily for 14 days.
  Interventions: Drug: Bifidobacterium Infants plus Enterococcus Feacium plus Lactobacillus Acidophilus
- Group 2 (Linex ® group) (Active Comparator): consists of 46 patients who will receive Amoxicillin 1 gm three times daily plus Lansoprazole 30 mg three times daily plus Linex ® capsule (which contains Bifidobacterium Infants, Enterococcus Feacium, and Lactobacillus Acidophilus) 1 capsule three times daily for 14 days.
  Interventions: Drug: Bifidobacterium Infants plus Enterococcus Feacium plus Lactobacillus Acidophilus

INTERVENTIONS:
Drug: Bifidobacterium Infants plus Enterococcus Feacium plus Lactobacillus Acidophilus — Bifidobacterium Infants, Enterococcus Feacium, and Lactobacillus Acidophilus combination will be given as one capsule three times daily for 14 days
  Other Names: linex

SUMMARY:
This study aims to investigate the possible safety and efficacy of probiotics (Bifidobacterium Infants, Enterococcus Feacium, and Lactobacillus Acidophilus) on the eradication rate of Helicobacter pylori and the incidence of adverse effects (AEs) of the concurrent rescue regimen in a patient with persistent H. Pylori infection.

DETAILED DESCRIPTION:
Over fifty percent of people worldwide are infected with the gram-negative bacteria Helicobacter pylori. This bacterial infection results in chronic gastritis and is a known risk factor for the development of gastric cancer, the second most lethal disease globally and the fourth most prevalent cancer overall.

The incidence and prevalence rates of H. Pylori in Egypt are relatively high, according to a previous study that covered the Delta region of the country, low socioeconomic status, poor sanitation, and fecal contamination of food or water are all associated with a high H. pylori prevalence.

During the COVID-19 pandemic, antibiotic resistance has been significantly rising in several countries as a result of the multiple preventative and treatment procedures being used to manage bacterial pneumonia that co-exist with the COVID-19 virus. The incidence of bacterial antibiotic resistance varies locally and seems to be changing over time in various regions, and as a result, the rate of H. pylori eradication worldwide is declining.

In about 20% of patients, an initial attempt to eradicate H. pylori fails, leaving them with a persistent infection so, it is crucial to choose medications carefully because H. pylori resistance to previously successful antibiotic treatments is on the rise. Poor nutrition, uncooperative patients, a high bacterial load in the stomach, internalization of germs, gastric acidity, gene polymorphisms, antimicrobial washout, and, most critically, antibiotic resistance are some of the variables that contribute to the failure of H. pylori eradication, severe consequence, and persistent infection.

The initial treatment plan, the usage of different antibiotics, and the existence of drug allergies should all be taken into consideration when choosing antibiotic therapy for patients with persistent H. pylori infection. It is normally advised to avoid using antibiotics included in the initial regimen. Amoxicillin can be taken again, though, as resistance seldom arises.

According to the 2022 Maastricht VI/Florence consensus report for Management of H. pylori infection, a PPI-Amoxicillin high-dose might be an option as rescue therapy, as it overcomes the issue of clarithromycin, metronidazole, or levofloxacin resistance. Fortunately, amoxicillin resistance prevalence as a beta-lactamase antibiotic has remained low and some studies reported 2% resistance in countries.

A Meta-analysis included 4 RCTs administering PPI-Amoxicillin dual therapy had an unacceptable eradication rate of 73%, which is comparable to other recommended therapies. While another recent RCT aimed to evaluate the effectiveness, compliance, and safety of High-Dose Dual Therapy (HDDT) in the management of H. pylori infection as ﬁrst-line treatment and as rescue therapy, revealed that the effectiveness of HDDT was below 70% in all scenarios (both ﬁrst-line and rescue treatment) and specifically was 48.4 % per protocol in patients who have been treated with HDDT as rescue treatment for 14 days.

However, further Studies are still needed to identify the effectiveness of this regimen, especially with the high antimicrobial resistance during COVID-19.

Probiotics are frequently thought to help with H. pylori eradication and lessen adverse effects caused by standard treatment. Inhibiting H. pylori colonization and adhesion which is important in determining the outcome of H. pylori-related diseases, decreasing inflammation brought on by H. pylori, modulating the immunological responses of H. pylori, lowering the frequency of side effects, and consequently increasing compliance were a handful possible mechanisms.

Probiotics may affect host immune responses by interacting with epithelial cells and regulating the release of anti-inflammatory cytokines brought on by H. pylori, which may lessen stomach activity and inflammation. The cytokine response first manifests as the production of IL-8, which causes neutrophils and monocytes to migrate to the mucus. As a result, IL-4, IL-5, IL-6, and INF- cytokines are produced by these activated monocytes and dendritic cells.

By creating organic acids, hydrogen peroxide, carbon dioxide, and other antimicrobial chemicals, probiotics like lactic acid bacteria (LAB) and Bifidobacterium may generally suppress other infections. As an add-on, Some Lactobacillus species generate bacteriocin-related antibacterial substances that may have antibacterial properties. In comparison to other strains, certain bacteriocins have more potent antibacterial action against H. pylori. Bacteriocin-like compound with an antagonistic effect against H. pylori was generated by Enterococcus faecium TM39 which inhibited the development of H. pylori.

Previous studies have examined the efficacy and safety of some types of probiotics in helicobacter pylori eradication therapy. But there is no study yet that has examined the efficacy and safety of Lactobacillus, Enterococcus- and Bifidobacterium-containing Probiotic combination on the eradication rate in persistent H. Pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with persistent H. pylori infection of both sexes aged ≥ 18 years old years whose infection was previously confirmed by endoscopy and pathology and experienced ≥ 2 previous treatment failures.

Exclusion Criteria:

* Patients with penicillin allergy.

  * Patients who have severe renal or hepatic disease.
  * Patients who have severe cardiovascular, endocrinological or pulmonary disease.
  * Patients with neoplastic diseases in the 5 years previous to recruitment.
  * Patients with neurological or psychiatric pathology.
  * Pregnant and/or lactating females
  * Patients with a history of allergic reactions to any medications used in the study.
  * Patients with a history of taking proton pump inhibitors, H2 antagonists, bismuth, or antibiotics (amoxicillin, metronidazole, clarithromycin) in the previous 2 weeks.
  * Patients on N-acetylcysteine
  * Patients on drug or alcohol abuse in the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
eradication of H. Pylori infection | 4-6 weeks after completion of therapy
  the eradication of H. Pylori infection which will be measured by stool antigen test, 4-6 weeks after completion of therapy. Eradication failure is defined as a positive result 4-6 weeks after completing therapy

SECONDARY OUTCOMES:
The improvement in Glasgow dyspepsia questionnaire | at baseline and after 8 weeks
  The Glasgow dyspepsia questionnaire is an eight-item self-reported dyspepsia specific questionnaire. It yields a global score that ranges from 0 to 20 and higher scores indicate more severe dyspepsia.
  It will be used for assessing the response to treatment in patients with dyspepsia at baseline and after 8 weeks.
Decrease incidence of adverse drug reactions | at day 7, 14, 21, and 28 after dug administration
  Side effects will be described as symptoms occurring after ingestion of medication and will be assessed at 7, 14, 21, and 28 days by telephone calls and through direct meetings.
change in Serum Pepsinogen (PG) I/II ratio | at baseline and after 8 weeks
  the percentage changes in Serum Pepsinogen (PG) I/II ratio) we will be evaluated for determining the success of eradication therapy for H. pylori. A significant increase in the pepsinogen I/II ratio is an indicator of successful Helicobacter pylori eradication.
change in Serum Interleukin 8 (IL-8) | at baseline and after 8 weeks
  Change in Serum Interleukin 8 (IL-8) will be measured at baseline and after 8 weeks. A significant increase in serum IL-8 level is an indicator of successful Helicobacter pylori eradication because when Tissue IL-8 levels decrease toward baseline levels following eradication of H pylori infection by antibiotic therapy, the serum IL-8 levels increase.

CONTACTS AND LOCATIONS:
Overall Officials: Noura Elsaka, Principal Investigator — Tanta University; Mohamed Abd El-Moaty, Professor, Study Chair — Zagazig University; Sahar Hegazy, Professor, Study Director — Tanta University
Locations (1):
- Faculty of medicine- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No